CLINICAL TRIAL: NCT03164590
Title: Effects of Local Wound Infiltration With Ketamine Versus Dexmedetomidine Added to Bupivacaine on Inflammatory Cytokines Response After Total Abdominal Hysterectomy
Brief Title: Effects of Wound Infiltration With Ketamine Versus Dexmedetomidine Added to Bupivacaine on Cytokines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia ,ICU and pain releif, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 388
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-01

CONDITIONS: Endometrial Adenocarcinoma
MeSH Terms: interventions — Ketamine; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ketamine (Active Comparator)
  Interventions: Drug: Ketamine
- dexmedetomidine (Active Comparator)
  Interventions: Drug: dexmedetomidine
- bupivacaine (Placebo Comparator)
  Interventions: Drug: Ketamine; Drug: dexmedetomidine; Drug: bupivacaine

INTERVENTIONS:
Drug: Ketamine — patients receive local anesthetic wound infiltration with 1 mg /kg ketamine
  Arms: bupivacaine; ketamine
Drug: dexmedetomidine — patients receive local anesthetic wound infiltration with 1µg/kg dexmedetomidine
  Arms: bupivacaine; dexmedetomidine
Drug: bupivacaine — patients receive local anesthetic wound infiltration with bupivacaine 0.5 % diluted in 20 ml saline
  Arms: bupivacaine

SUMMARY:
This study aims to compare the effects of local wound infiltration with ketamine versus dexmedetomidine when added to bupivacaine on inflammatory cytokine response after total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* age range (18-60) years,
* weight (50- 90) kg

Exclusion Criteria:

* allergy to study drugs
* significant cardiac disease
* respiratory disease
* renal disease
* hepatic disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
severity of pain at rest and on coughing | 24 hours
  severity of pain at rest and on coughing will be assessed using a 10-cm Visual Analog Scale (0 = no pain and 10 = worst imaginable pain)

SECONDARY OUTCOMES:
sedation | 24 hours
  sedation by using sedation score

CONTACTS AND LOCATIONS:
Overall Officials: fatma el sherif, MD, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- South Egypt Cancer instIitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No